CLINICAL TRIAL: NCT06064357
Title: Comparison of Massage Therapy and Tissue Flossing Technique in Children With Diplegic Cerebral Palsy
Brief Title: Comparison of Massage Therapy and Tissue Flossing Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEMRA SHAH REC/PT/01591
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Spastic Diplegia Cerebral Palsy
Keywords: Massage Therapy, Tissue Flossing, Diplegia cerebral palsy,
MeSH Terms: conditions — Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Intervention Model Description: Transverse friction massage at Rectus femoris, hip adductors, hamstring, and calf of both lower limbs.Applied time is 30 seconds, 3 sets with 10 seconds rest interval after that massage will be performed on next group of muscle.4 time / week for 6 weeks.
  Conventional physical therapy program included application hot pack for 15 minutes, and Bobath treatment followed by stretching of calf muscles (10 repetitions with at least 8 seconds hold) 4 times / week for 6 weeks.
  Tissue floss band will be applied on Rectus femoris, hip adductors, calf and hamstring of both lower limbs. Floss band will be wrap around the particular muscle from distal to proximal direction with 25 % stretch and 50% overlap and then 10 Reps of rom will be actively performed and then the rest interval is 2 mints. 4 sessions / week for 6 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transverese friction massage + Conventional Physio Therapy (Experimental): Transverse friction massage: Transverse friction massage at Rectus femoris, hip adductors, hamstring, and calf muscle on both lower limbs. TFM on each group of muscle for 30 seconds, 3 sets with 10 seconds rest interval after that massage will be performed on next group of muscle.4 session per week lasting for 6 weeks.
  Conventional Therapy:
  Conventional physical therapy program included application hot pack for 15 minutes, and Bobath treatment followed by stretching of calf muscles (10 repetitions with at least 8 seconds hold) 4 times a week lasting for 6 weeks
  Interventions: Other: Transverese friction massage and tissue floss technique
- Tissue flossing technique + Conventional Physio Therapy (Experimental): Tissue floss bands: These band will be applied on Rectus femoris, hip adductors, calf muscle and hamstring muscle of both lower limbs. Floss band will be wrap around the particular group of muscle from distal to proximal direction with 25 % stretch and 50% overlap a few inches below and few inches above the area and then 10 Reps of rom will be actively performed by the participants and then after 10 Reps remove the band and the rest interval is 2 mint after that next group of muscle will be wrap. 4 sessions per week lasting for 6 weeks.
  Conventional Therapy: Conventional physical therapy program included application hot pack for 15 minutes, and Bobath treatment followed by stretching of calf muscles (10 repetitions with at least 8 seconds hold) 4 times a week lasting for 6 weeks.
  Interventions: Other: Transverese friction massage and tissue floss technique

INTERVENTIONS:
Other: Transverese friction massage and tissue floss technique — Transverse friction massage at Rectus femoris, hip adductors, hamstring, and calf of both lower limbs. TFM on each group of muscle for 30 seconds, 3 sets with 10 seconds rest interval.4 session / week for 6 weeks.
  Tissue floss band will be applied on Rectus femoris, hip adductors, calf and hamstring of both lower limbs. Floss band will be wrap around the particular group of muscle from distal to proximal direction with 25 % stretch and 50% overlap and then 10 Reps of rom will be performed the rest interval is 2 mint. 4 sessions / week for 6 weeks.
  Conventional physical therapy program included application hot pack for 15 minutes, and Bobath treatment followed by stretching of calf (10 repetitions with at least 8 seconds hold) 4 times / week for 6 weeks.

SUMMARY:
The purpose of the study is to compare massage therapy with tissue flossing technique in children with diplegic cerebral palsy. A randomized control trial would be conducted at helping hand for relief and development Quetta. The sample size is 56 calculated through G power. The participants would be divided into two interventional groups each having 28 participants. The study duration would be six weeks. Sampling technique applied would be convenient sampling for recruitment and group randomization via using envelop method. Tools used in this study are Goniometer, muscle length test and Functional Mobility scale. Data would be collected before and after 6 weeks of the application of interventions. Data analyzed through SPSS version 23.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a syndrome of motor impairments characterized by non-progressive disturbances taking place in developing fetal and infant brain(1). The most prevalent motor disability in children, CP affects 2 to 3 out of every 1,000 live births. The most prevalent type of CP, spastic CP account for about 80% , especially spastic diplegic, accounts for between 50% and 60% of all cases(2).The term "cerebral paralysis "was used for the ﬁrst time in 1861, by the English orthopedic surgeon named William Little (3). There are four categories of risk factors for CP: pre-conception, prenatal, perinatal, and postnatal(3, 4). Traditionally, CP has been categorized according to the type of movement dysfunction and anatomical distribution. Spastic, dyskinetic, hypotonic, ataxic, and mixed kinds of movement are among the patterns of movement. Spastic movement is the most prevalent, with dyskinetic, ataxic, or hypotonic movement patterns making up the minority of cases(5). Hemiplegic, diplegic, and quadriplegic made up the anatomic distribution. Only one side of the body is affected in hemiplegic CP, and the upper extremities often show the greatest deficits. Lower extremities are more commonly affected in Diplegic CP than upper extremities. The axial and appendicular skeletons are both affected in Quadra plegic cerebral palsy, which affects the entire body (6).

Damage to the brain occurs in CP patients, most frequently in the region of the brain that regulates muscle tone and limb movement. As a result, the brain is powerless to control how flexible a muscle should be. The spinal cord is dominated by the command from the muscle, which causes the muscle to become too tight or spastic(7). Periventricular leukomalacia (PVL), the most prevalent abnormality on neuroimaging, is a white matter anomaly located close to the lateral ventricle. Children with PVL often exhibit spastic diplegia because the corticospinal tract fibers to the lower limbs are medial to those of the upper extremities in the periventricular white matter(3, 8).CP child are diagnosed on the basis of history and physical examination(2). Muscle stiffness and heightened reflexes are side effects of cerebral palsy, which affects mobility and coordination. Either too loose or too rigid a muscle tone. Walking difficulty, such as walking on one's toes or crossing one's knees like a scissor. Inability to use fine motor abilities. Balance and muscle coordination are noticeably absent. Tremors and jerky involuntary movement also present in children with athetoid CP(3,9).Spasticity causes irregular movements in the muscles and joints of the extremities and is particularly damaging to growing youngsters. Any muscle group in the body might be affected by spasticity. Hip flexion, adduction of the thighs, knee flexion, equinovarus foot posture, and hyperextension of the big toe are the effects on the lower limbs.(7). In spastic diplegia the most commonly effected lower limb muscles are gastrocnemius, soleus, adductors, hamstrings, psoas and rectus femoris(2).

The treatment of a child with CP requires a multidisciplinary approach(7). Physiotherapy intervention included static and dynamic weight bearing exercises balance training, weight bearing exercises, sustained stretching exercises, Roods approach, Bobath technique, exercises on Swiss ball, orthosis, and proper home exercise program(10).Massage is one of the oldest and most widely used treatments in complementary and alternative medicine, with more than 75 forms of it practiced today(2).Massage has positive effects on muscle tone disorder(11, 12).Mocgregor et al conducted a study in this Transverse-friction massage was applied to the calf muscles of patients with spastic diplegia. They hypothesized that this resets sarcomere length(8).Tissue flossing was first proposed by Starrett and Cordoza (2015), who claimed that it can lessen discomfort from various diseases or injuries, increase range of motion, and/or improve performance (such as strength or leaping performance(13). The flexibility of muscles can be greatly increased with Floss Band intervention(14, 15).

Generally, muscles of children with CP lack muscular flexibility. Muscular stiffness results from an increase in muscular tone. Due to muscular stiffness, it was impossible to stretch the muscle properly, which led to the creation of contractures, reduced range of motion (ROM), and restricted mobility. Muscular flexibility is a basic element for muscular action and important milestone in the rehabilitation program for children with CP.

Treatment options provided to improve muscles flexibility, rang of motion and mobility of children with CP must not be limited to invasive methods which are also financially expensive. The Tissue flossing is a novice, non-invasive method that depend on an easily held, safe, cheap and light weighted. The use of tissue flossing is becoming a popular strategy in rehabilitation program. However the literature on floss band effectiveness in children with Cp remain sparse. Previously studies have been conducted that support the role of tissue flossing in athletes and in individuals with various musculoskeletal injuries. However its role particularly in CP patients is unavailable. In this research we have incorporated this technique to determine its effects in cerebral palsy children. Therefore, the purpose of this study is to do comparison between transverse friction massage with tissue flossing technique and examine the effects on range of motion, muscular flexibility, and mobility in children with diplegic CP.

ELIGIBILITY:
Inclusion Criteria:

Participants falling in this category would be recruited into the study.

* Both genders (male and female).
* Age between 12 - 15 years.
* Diagnosed patients of spastic diplegic cerebral palsy.
* Muscle tone between (1 and 1+) according to modified Ashworth scale.
* Gross motor function classification system level will be from I to IV.
* Children who has communication skills (according to communication function classification system, level I - III).

Exclusion Criteria:

Participants falling in this category would be excluded from the study.

* Previous Fracture/Trauma of lower limb less than six month prior to the study.
* Soft tissue injury of lower limb less than six month prior to the study.
* History of any surgical intervention for the management of spasticity or any orthopedic surgery of lower limb.
* Any therapeutic intervention for the management of spasticity i-e (botulinum injections, ITB and drugs) less than six month prior to the study.
* Children with multiple disabilities.
* Seizure.
* Latex allergy.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-01-05 (Estimated); Study Completion 2024-01-28 (Estimated)

PRIMARY OUTCOMES:
Goniometery | Base Line measurement before start of treatment and post 6th Week
  It is an instrument that measures the available range of motion at a joint. It will used to determine range of motion of hip, knee and ankle joint (16).
Muscle length test | Base Line measurement before start of treatment and post 6th Week
  Muscle length test of rectus femoris, hip adductors, hamstring, gastrocnemius and soleus will be performed to determined muscular flexibility (17).
Functional mobility scale | Base Line measurement before start of treatment and post 6th Week
  It is an instrument that measures the available range of motion at a joint. Functional mobility scale will be used to determined mobility (18).

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MScNMPT, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand For Relief and Development Quetta, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monokwane B, Johnson A, Gambrah-Sampaney C, Khurana E, Baier J, Baranov E, Westmoreland KD, Mazhani L, Steenhoff AP, Bearden DR. Risk Factors for Cerebral Palsy in Children in Botswana. Pediatr Neurol. 2017 Dec;77:73-77. doi: 10.1016/j.pediatrneurol.2017.07.014. Epub 2017 Aug 3. PMID 29074060
- [Background] Rasool F, Memon AR, Kiyani MM, Sajjad AG. The effect of deep cross friction massage on spasticity of children with cerebral palsy: A double-blind randomised controlled trial. J Pak Med Assoc. 2017 Jan;67(1):87-91. PMID 28065961
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Yuan J, Wang J, Ma J, Zhu D, Zhang Z, Li J. Paediatric cerebral palsy prevalence and high-risk factors in Henan province, Central China. J Rehabil Med. 2019 Jan 1;51(1):47-53. doi: 10.2340/16501977-2486. PMID 30299526
- [Background] Lee H, Kim EK, Son DB, Hwang Y, Kim JS, Lim SH, Sul B, Hong BY. The Role of Regular Physical Therapy on Spasticity in Children With Cerebral Palsy. Ann Rehabil Med. 2019 Jun;43(3):289-296. doi: 10.5535/arm.2019.43.3.289. Epub 2019 Jun 28. PMID 31311250
- [Background] Pavone P, Gulizia C, Le Pira A, Greco F, Parisi P, Di Cara G, Falsaperla R, Lubrano R, Minardi C, Spalice A, Ruggieri M. Cerebral Palsy and Epilepsy in Children: Clinical Perspectives on a Common Comorbidity. Children (Basel). 2020 Dec 31;8(1):16. doi: 10.3390/children8010016. PMID 33396243
- [Background] Dimitrijević L, Čolović H, Spalević M, Stanković A, Zlatanović D, Cvetković B. Assessment and treatment of spasticity in children with cerebral palsy. Acta Facultatis Medicae Naissensis. 2014;31(3):163-9.
- [Background] Macgregor R, Campbell R, Gladden MH, Tennant N, Young D. Effects of massage on the mechanical behaviour of muscles in adolescents with spastic diplegia: a pilot study. Dev Med Child Neurol. 2007 Mar;49(3):187-91. doi: 10.1111/j.1469-8749.2007.00187.x. PMID 17355474
- [Background] Raut A, Risaldar P, Naqvi WM, Wane M, Sahu A. Case report of a spastic diplegic cerebral palsy patient: Clinical decision making in physical therapy. 5. Medical Science. 2020;24(103):1809-13.
- [Background] Field T. Pediatric Massage Therapy Research: A Narrative Review. Children (Basel). 2019 Jun 6;6(6):78. doi: 10.3390/children6060078. PMID 31174382
- [Background] Bingöl H, Akaras E, Kocaman H. The effects of massage therapy on symptoms related cerebral palsy in children with cerebral palsy: A systematic review. Journal of Clinical Medicine of Kazakhstan. 2020;4(58):6-14.
- [Background] Konrad A, Mocnik R, Nakamura M. Effects of Tissue Flossing on the Healthy and Impaired Musculoskeletal System: A Scoping Review. Front Physiol. 2021 May 21;12:666129. doi: 10.3389/fphys.2021.666129. eCollection 2021. PMID 34093228
- [Background] Chang N-J, Hung W-C, Lee C-L, Chang W-D, Wu B-H. Effects of a single session of floss band intervention on flexibility of thigh, knee joint proprioception, muscle force output, and dynamic balance in young adults. Applied Sciences. 2021;11(24):12052.
- [Background] Stuberg WA, Fuchs RH, Miedaner JA. Reliability of goniometric measurements of children with cerebral palsy. Dev Med Child Neurol. 1988 Oct;30(5):657-66. doi: 10.1111/j.1469-8749.1988.tb04805.x. PMID 3229564
- [Background] Kaneda H, Takahira N, Tsuda K, Tozaki K, Sakai K, Kudo S, et al. The effects of tissue flossing and static stretching on gastrocnemius exertion and flexibility. Isokinetics and Exercise Science. 2020;28(2):205-13.
- [Background] Pawar A, Phansopkar P, Gachake A, Mandhane K, Jain R, Vaidya S. A review on impact of lower extremity muscle Length. J Pharm Res Int. 2021;33(35A):158-64.
- [Background] Ammann-Reiffer C, Bastiaenen CHG, Van Hedel HJA. Measuring change in gait performance of children with motor disorders: assessing the Functional Mobility Scale and the Gillette Functional Assessment Questionnaire walking scale. Dev Med Child Neurol. 2019 Jun;61(6):717-724. doi: 10.1111/dmcn.14071. Epub 2018 Oct 19. PMID 30341775